CLINICAL TRIAL: NCT02125994
Title: Comparison of the Effect of Ropivacaine 0.5% vs 0.375% on the Autonomous Nervous System During Shoulder Surgery in Beach Chair Position
Brief Title: Effect of 0.5% vs 0.375% Ropivacaine on Autonomous Nervous System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Larissa University Hospital (Other)
Responsible Party: Principal Investigator, Marina Simaioforidou, Anesthesiologist, Larissa University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Shoulder 0.5 vs 0.375
Record Dates: First submitted 2014-04-27; First posted 2014-04-29 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Shoulder Surgery; Interscalene Nerve Block; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine 0.5% (Active Comparator): Ultrasound guided Intercalene nerve block with ropivacaine 0.5 %
  Interventions: Procedure: Interscalene nerve block
- Ropivacaine 0.375 % (Active Comparator): Ultrasound guided Intercalene nerve block with ropivacaine 0.375 %
  Interventions: Procedure: Interscalene nerve block

INTERVENTIONS:
Procedure: Interscalene nerve block

SUMMARY:
It is established that the local anesthetic that is administered during an interscalene block affects the autonomic outflow to the heart. This is very well seen during shoulder surgery when the patient is positioned in beach chair pasition.

The investigators want to study the different effect of the two concentrations (0.5% and 0.375%) of ropivacaine on the autonomic nervous system through blood pressure and heart rate measurements.

ELIGIBILITY:
Inclusion Criteria:

* Elective shoulder surgery
* Age 18- 80 years old
* ASA I - IV
* Beach chair position

Exclusion Criteria:

* Coagulopathy disorders
* Infection at the puncture site for the interscalene block
* Neurological deficit on the side to be operated
* Allergy to local anesthetics
* Psychiatric disorders
* Patient's refusal
* Problems with patient communication
* Failure of the interscalene block

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Blood pressure fluctuations | Completion of the surgery

SECONDARY OUTCOMES:
Heart rate fluctuations | Completion of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marina Simaioforidou, Medicine, Study Director — Private Clinic of Larissa "Asklipeiio"; Metaxia Bareka, Medicine, Principal Investigator — University Hospital of Larisa; George Basdekis, Medicine, Study Chair — Private Clinic of Larissa "Asklipeiio"; Konstantinos Bargiotas, Medicine, Study Chair — Larissa University Hospital; Sokrates Varitimidis, Medicine, Study Chair — Larissa University Hospital; Aristeidis Zibis, Medicine, Study Chair — Private Clinic of Larissa "Asklipeiio"; Konstantinos Alexiou, Medicine, Study Chair — Larissa University Hospital
Locations (1):
- Private Clinic of Larissa "Asklipeiio", Larissa, Larissa, Greece